CLINICAL TRIAL: NCT02876302
Title: Phase II Study Of Combination Ruxolitinib (INCB018424) With Preoperative Chemotherapy For Triple Negative Inflammatory Breast Cancer
Brief Title: Study Of Ruxolitinib (INCB018424) With Preoperative Chemotherapy For Triple Negative Inflammatory Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Filipa Lynce, MD, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-151
Record Dates: First submitted 2016-08-09; First posted 2016-08-23 (Estimated); Results first posted 2024-04-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Breast Cancer (IBC)
Keywords: Inflammatory Breast Cancer; Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — ruxolitinib; Paclitaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Paclitaxel (12weeks) (Experimental): Paclitaxel is administered weekly followed by standard Doxorubicin and Dyclophosphamide (AC) given every 2 weeks for 4 cycles preoperatively
  * 16 patients will be randomized from the Run-In 7 days of Ruxolitinib
  * The drug will be administered at a pre-determine dosage
  Interventions: Drug: Ruxolitinib; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide
- Ruxolitinib with Paclitaxel (12weeks) (Experimental): Paclitaxel is administered with daily Ruxolitinib, followed by standard Doxorubicin and Cyclophosphamide (AC) given every 2 weeks for 4 cycles preoperatively
  * 16 patients will be randomized from the Run-In 7 days of Ruxolitinib
  * The drug will be administered at a pre-determine dosage
  Interventions: Drug: Ruxolitinib; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide
- Ruxolitinib and Paclitaxel (12weeks) (Experimental): Paclitaxel is administered with daily Ruxolitinib, followed by standard Doxorubicin and Cyclophosphamide (AC) given every 2 weeks for 4 cycles preoperatively
  * 32 patients will be randomized from the Run-In 7 days of Ruxolitinib + Paclitaxel
  * The drug will be administered at a pre-determine dosage
  Interventions: Drug: Ruxolitinib; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Ruxolitinib — 15 or 20 mg, twice daily by mouth. The run-in part of ruxolitinib lasts 7 days; The treatment of ruxolitinib part lasts 12 weeks.
  Other Names: Jakafi
Drug: Paclitaxel — 80 mg/m2, IV (in the vein) weekly for 12 weeks.
  Other Names: Taxol
Drug: Doxorubicin — 60 mg/m2, IV (in the vein) every 14 days for 4 doses.
  Other Names: Adriamycin
Drug: Cyclophosphamide — 600 mg/m2, IV (in the vein) every 14 days for 4 doses.
  Other Names: Cytoxan

SUMMARY:
This research study is studying Ruxolitinib as possible treatment for Inflammatory Breast Cancer (IBC).

The Following drugs will be use in combination with Ruxolinitinib.

* Paclitaxel (also called Taxol)
* Doxorubicin also called Adriamycin
* Cyclophosphamide, also called Cytoxan

DETAILED DESCRIPTION:
This is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (U.S. Food and Drug Administration) has not approved Ruxolitinib for Inflammatory Breast Cancer (IBC), but is has been approved for other uses.

Ruxolitinib is a newly discovered drug that has been shown to block a pathway (called the IL6/JAK/Stat pathway) that may be important in cancer, including triple negative inflammatory breast cancer. Ruxolitinib brings proteins groups together, which can result in gene (DNA) changes. These DNA changes may stop cancer cells from growing.

Paclitaxel (also called Taxol), Doxorubicin and Cyclophosphamide (also called Adriamycin and Cytoxan, ("AC")) are drugs FDA approved for breast cancer patients. They have been shown to result in death of cancer cells when given as preoperative treatment of women with inflammatory breast cancer (IBC). Laboratory studies have shown that Ruxolitinib may make Paclitaxel more effective.

In this research study, the investigators are evaluating Ruxolitinib in combination with Paclitaxel followed by the standard chemotherapy, AC. Researchers will also evaluate how the IL6/JAK/Stat pathway is affected by this combination of drugs by studying biopsies and surgical specimens.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed invasive breast cancer. All histologic subtypes are eligible.
* Patients must have known ER, PR, and HER2 status defined as triple-negative breast cancer (TNBC), defined as:

  --ER and PR <10% by immunohistochemistry, and HER2-negative ( as per ASCO/CAP guidelines, defined as IHC 0 or 1+, or FISH ratio <2.0 or HER2 copy number <6.0).
* Patients must have the clinical diagnosis of inflammatory breast cancer, involving an intact breast.
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of ruxolitinib in participants <18 years of age, children are excluded from this study.
* ECOG performance status 0 or 1.
* Participants must have normal organ and marrow function as defined below:

  * Leukocytes ≥ 3,000/mm3
  * Absolute neutrophil count ≥ 1,500/mm3
  * Platelets ≥ 100,000/mm3
  * Bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
  * AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal
  * Creatinine ≤1.5 x institutional upper limit of normal OR creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
* Patients with evidence of extensive nodal involvement are allowed. Extensive nodal involvement is defined as metastatic disease involving any nodal region outside of the involved breast.
* Patients with minimal metastatic disease involvement in bone or viscera are allowed. Minimal metastatic disease is defined as: evidence of metastatic involvement as demonstrated by imaging only, not amenable to biopsy confirmation.
* Both men and women are allowed.
* The effects of ruxolitinib on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry until completion of chemotherapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* LVEF > 50% calculated by echocardiogram (ECHO) or MUGA
* Patients may have bilateral breast cancer so long as one breast meets criteria for inflammatory breast cancer, and neither breast cancer has received prior therapy

Exclusion Criteria:

* Participants may not be receiving any other investigational agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib.
* Participants receiving any medications or substances that are potent inhibitors of CYP3A4, including grapefruit juice are ineligible. Participants receiving fluconazole are also ineligible. (Please refer to Appendix B for the full list of potent inhibitors and washout periods).
* Chronic corticosteroid use in excess of the equivalent of prednisone 10 mg once daily.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because paclitaxel, doxorubicin, and cyclophosphamide have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated on study. These potential risks may also apply to other agents used in this study.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Known HIV-positive individuals on combination antiretroviral therapy are eligible so long as they meet all other criteria. Known HIV-positive individuals who are not on combination antiretroviral therapy are not eligible because these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Clinically significant malabsorption syndrome.
* Patients may not have received paclitaxel, doxorubicin, or cyclophosphamide as anti-neoplastic therapy.
* Patients with prior radiation to the affected breast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Filipa Lynce, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lynce F, Stevens LE, Li Z, Brock JE, Gulvady A, Huang Y, Nakhlis F, Patel A, Force JM, Haddad TC, Ueno N, Stearns V, Wolff AC, Clark AS, Bellon JR, Richardson ET, Balko JM, Krop IE, Winer EP, Lange P, Hwang ES, King TA, Tolaney SM, Thompson A, Gupta GP, Mittendorf EA, Regan MM, Overmoyer B, Polyak K. TBCRC 039: a phase II study of preoperative ruxolitinib with or without paclitaxel for triple-negative inflammatory breast cancer. Breast Cancer Res. 2024 Jan 31;26(1):20. doi: 10.1186/s13058-024-01774-0. PMID 38297352

RESULTS

PARTICIPANT FLOW:
Groups:
- Ruxolitinib Alone First: Patients (n=11) receiving ruxolitinib alone (15 mg or 20mg orally, depending on initial platelet count) given in the run-in phase for 7 days.
- Ruxolitinib Plus Paclitaxel First: Patients (n=12) receive ruxolitinib (15 mg orally) twice daily for 7 days in combination with one dose of paclitaxel (80 mg/m2; administered on day 1, denoted Cycle 0, Day 1) in the run-in phase for 7 days.
Period: Run-In Treatment Phase
Arm/Group | Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel First
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0
Period: Neoadjuvant Treatment Phase
Arm/Group | Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel First
Started | 11 | 12
Treated with neoadjuvant paclitaxel Only | 6 | 0
Treated with neoadjuvant ruxolitinib and paclitaxel | 5 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treatment-naïve patients received a 7-day run-in window of ruxolitinib alone or ruxolitinib plus paclitaxel. The primary endpoint objective was the percent of pSTAT3-positive pre-window phase tumors that became pSTAT3-negative. (After the window phase, those who received ruxolitinib alone proceeded to neoadjuvant therapy with either ruxolitinib plus paclitaxel or paclitaxel alone for 12 weeks; those who had received ruxolitinib plus paclitaxel continued treatment for 12 weeks.
Groups:
- Ruxolitinib Alone First: Patients (n=11) receiving ruxolitinib alone (15 mg or 20mg orally, depending on initial platelet count) given in the run-in treatment phase for 7 days.
- Ruxolitinib Plus Paclitaxel First: Patients (n=12) receive ruxolitinib (15 mg orally) twice daily for 7 days in combination with one dose of paclitaxel (80 mg/m2; administered on day 1, denoted Cycle 0, Day 1) in the run-in treatment phase for 7 days.
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel First | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Median Age, Window Phase | 54 [51 to 68] | 47 [41 to 64] | 53 [41 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 12 | 22
  Black or African American | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23
Clinical N stage [Count of Participants; unit: Participants] — According to the American Cancer Society, the N category can be assigned a letter or a number, where N0 means nearby lymph nodes do not contain cancer and the higher the number after the N (such as N1, N2, or N3), the greater the cancer spread to nearby lymph nodes.
  Participants
    Unknown | 1 | 0 | 1
    cN0 | 0 | 1 | 1
    cN1 | 10 | 5 | 15
    cN2 | 0 | 2 | 2
    cN3 | 0 | 4 | 4
M stage [Count of Participants; unit: Participants] — According to the American Cancer Society, the M stage is an indicator for metastasis, where M0 indicates that no distant cancer spread has been found and M1 indicates that distant spread to distant organs or tissues is present.
  Participants
    Unknown | 1 | 1 | 2
    M0 | 9 | 11 | 20
    M1 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Biologic Response To 7-Day Run-In Window Phase Treatment of Ruxolitinib Alone or Ruxolitinib Plus Paclitaxel
Description: Biologic response to 7-day run-in phase treatment, defined as a change in phosphorylated STAT3 (pSTAT3) expression from moderate/high positive (pSTAT3-positive) in pre-run-in phase sample to negative or weakly positive/equivocal (pSTAT3-negative) in post-run-in samples. pSTAT3 status was determined by evaluating the percent positive cells and the strength of staining (weak vs. strong/moderate) in relation to positive and negative controls. A T-score was calculated based on percent-stained cells and intensity of staining and interpreted as follows: Scores 0-4 are negative/weakly positive (pStat3 negative) and 5-8 are moderate/high positive (pStat3 positive). Hence, pStat3 negative indicates a biologic response or a decrease in pSTAT3 levels.
Time Frame: 7 days
Population: A total of 23 patients were enrolled across 4 centers from January 24, 2018, to February 5, 2021. During the window phase of the trial, 11 patients received 7 days of ruxolitinib and 12 received ruxolitinib plus paclitaxel. Among 23 patients, 20 had baseline biopsy samples stained.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel First
Number analyzed (Participants) | 11 | 12
Participants
  pStat3 negative | 2 | 3
  pStat3 positive | 9 | 6
  Baseline pStat3 status not available | 0 | 3

2. Secondary Outcome: Pathologic Complete Response Rate (pCR) After Preoperative Therapy
Description: Pathologic Complete Response rate (pCR) is defined as the absence of invasive carcinoma within the breast and axillary lymph nodes following preoperative therapy.
Time Frame: 28 weeks
Population: Neoadjuvant treatment phase population including those who received single agent ruxolitinib during the window phase treatment and then proceeded to neoadjuvant therapy with daily ruxolitinib plus weekly paclitaxel for 12 weeks (n=5) and those patients who had received the combination of ruxolitinib plus paclitaxel during the window phase continued to receive it for a total of 12 weeks (n=12).
Measure: Count of Participants; unit: Participants
Groups:
- Paclitaxel Alone Given As Neoadjuvant Therapy, After Ruxolitinib Alone First: Ruxolitinib alone (15 mg or 20 mg orally, depending on initial platelet count) is given in the run-in phase for 7 days. After the run-in phase, patients (n=6) who received ruxolitinib alone proceeded to neoadjuvant therapy with paclitaxel alone (80 mg/m2) for 12 weeks. Two weeks after the last dose of paclitaxel, all patients received neoadjuvant doxorubicin and cyclophosphamide every two weeks for four cycles.
- Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy: After the run-in phase, patients (n=5) receiving single agent ruxolitinib (15 mg or 20 mg orally, depending on initial platelet count) twice daily for seven days, proceeded to neoadjuvant therapy with ruxolitinib plus paclitaxel for 12 weeks in addition to patients (n=12) who had received the combination of ruxolitinib plus paclitaxel (15 mg orally) twice daily for seven days in combination with one dose of paclitaxel (80 mg/m2; administered on day 1, denoted Cycle 0, Day 1) in the run-in phase, continued to receive the combination of ruxolitinib plus paclitaxel for a total of 12 weeks. Two weeks after the last dose of paclitaxel, all patients received neoadjuvant doxorubicin and cyclophosphamide every two weeks for four cycles.
Arm/Group | Paclitaxel Alone Given As Neoadjuvant Therapy, After Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy
Number analyzed (Participants) | 6 | 17
Participants
  pCR in breast and lymph nodes - No | 5 | 16
  pCR in breast and lymph nodes - Yes | 1 | 1

3. Secondary Outcome: Assess Change in STAT3 Gene Expression Following run-in Treatment
Description: Change of STAT3 gene expression between pretreatment and post-ruxolitinib run-in (after 7 days of ruxolitinib alone or with one dose of weekly paclitaxel) biopsy specimens. RNA-seq was performed on a subset of tumor pairs (n=4 per run-in treatment group). Enrichment analysis for JAK-STAT and IL-6 Hallmark signatures obtained a Gene Set Variation Analysis (GSVA) enrichment score as a measure of STAT3 gene expression. The GSVA enrichment score is a continuous unitless measure that summarizes joint expression of multiple genes into a single value. A positive value indicates greater, and a negative value a lesser, enrichment of pathway signatures; thus a negative pre- to post-runin change in the value indicates a decrease in the STAT3 expression after the treatment, and a positive values indicates increase in STAT3 expression after treatment.
Time Frame: 7 Days
Population: To assess global transcriptomic changes during treatment, RNA-seq was performed on paired pre- and post-run-in phase tumor biopsy samples (n=4 per run-in treatment group).
Measure: Mean (Standard Deviation); unit: GSVA enrichment score
Units Other Than Participants: Tumor pairs
Groups:
- Ruxolitinib Alone First: Patients receiving ruxolitinib alone (15 mg or 20mg orally, depending on initial platelet count) given in run-in phase for 7 days.
- Ruxolitinib Plus Paclitaxel First: Patients receive ruxolitinib (15 mg orally) twice daily for 7 days in combination with one dose of paclitaxel (80 mg/m2; administered on day 1, denoted Cycle 0, Day 1) in the run-in phase for 7 days.
Arm/Group | Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel First
Number analyzed (Participants) | 11 | 12
Number analyzed (Tumor pairs) | 4 | 4
GSVA enrichment score | -0.06 (0.23) | 0.01 (0.15)

4. Secondary Outcome: Determine Efficacy Defined as Disease-Free Survival (DFS)
Description: Disease-Free Survival (DFS) is defined as time of surgery, among the subset of patients who underwent surgery (n=21), until occurrence of recurrence, contralateral cancer, death attributable to any cause, second primary cancer other than breast. DFS was censored at date of last assessment.
Time Frame: 2 years
Population: Two patients whose disease progressed during neoadjuvant therapy did not have surgery; the other 21 patients proceeded to surgery and radiation therapy.
Measure: Count of Participants; unit: Participants
Groups:
- Paclitaxel Alone Given As Neoadjuvant Therapy, After Ruxolitinib Alone First: Ruxolitinib alone (15 mg or 20 mg orally, depending on initial platelet count) is given in the run-in phase for 7 days. After the run-in phase, patients (n=6) who received ruxolitinib alone proceeded to neoadjuvant therapy with paclitaxel alone (80 mg/m2) for 12 weeks. All patients subsequently received 4 cycles of doxorubicin plus cyclophosphamide prior to surgery.
- Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy: After the run-in phase, patients (n=5) receiving single agent ruxolitinib (15 mg or 20 mg orally, depending on initial platelet count) twice daily for seven days, proceeded to neoadjuvant therapy with ruxolitinib plus paclitaxel for 12 weeks in addition to patients (n=12) who had received the combination of ruxolitinib plus paclitaxel (15 mg orally) twice daily for seven days in combination with one dose of paclitaxel (80 mg/m2; administered on day 1, denoted Cycle 0, Day 1) in the run-in phase, continued to receive the combination of ruxolitinib plus paclitaxel for a total of 12 weeks. Subsequently 15 of 17 patients received 4 cycles of doxorubicin plus cyclophosphamide prior to having surgery; 2 of 17 patients had a progression of their disease during neoadjuvant therapy and hence did not proceed to surgery and radiation therapy.
Arm/Group | Paclitaxel Alone Given As Neoadjuvant Therapy, After Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy
Number analyzed (Participants) | 6 | 15
Participants
  DFS event - yes | 4 | 8
  DFS event - no | 2 | 7

5. Secondary Outcome: Determine Efficacy Defined as Time to Treatment Failure (TTF)
Description: The endpoint is now more commonly known as event-free survival (EFS). Defined as time of treatment initiation until occurrence of recurrence, contralateral cancer, death attributable to any cause, second primary cancer other than breast or occurrence of progressive disease during preoperative therapy or treatment of disease that is not surgically resectable; otherwise censored at last disease follow-up.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel Alone Given As Neoadjuvant Therapy, After Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy
Number analyzed (Participants) | 6 | 17
Participants
  EFS event - yes | 4 | 10
  EFS event - no | 2 | 7

6. Secondary Outcome: Determine Efficacy Defined as Overall Survival (OS)
Description: Overall survival (OS) is defined as time from surgery until death from any cause or from treatment initiation until death from any cause.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel Alone Given As Neoadjuvant Therapy, After Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy
Number analyzed (Participants) | 6 | 17
Participants
  OS event - yes | 3 | 5
  OS event - no | 3 | 12

7. Secondary Outcome: Assess Residual Cancer Burden (RCB) Differences After Preoperative Therapy
Description: Residual cancer burden (RCB) is a continuous variable (RCB0 through RCB-IV) derived from the primary tumor dimensions, cellularity of the tumor bed, and axillary nodal burden as described in Symmans et al, 2007; where RCB-0 equals pathologic complete response (pCR) and considered the best prognosis and RCB-IV is considered the worst prognosis.
Time Frame: 28 weeks
Population: Subset (n=15, patients allocated to ruxolitinib plus paclitaxel given as neoadjuvant therapy) of the overall patient population allocated to ruxolitinib plus paclitaxel given as neoadjuvant therapy (n=17) who had tumor samples at both baseline and 28 wk timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel Alone Given As Neoadjuvant Therapy, After Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy
Number analyzed (Participants) | 6 | 17
Participants
  RCB-0 (pCR) | 1 | 1
  RCB-I | 1 | 1
  RCB-II | 0 | 2
  RCB-III | 1 | 2
  RCB-IV | 3 | 9
  No surgery due to disease progression during neoadjuvant therapy | 0 | 2

8. Secondary Outcome: Changes in Interleukin 6 (IL-6) Plasma Levels During Treatment
Description: Elevations in interleukin (IL-6) and C-reactive protein (CRP) have been associated with worse clinical outcomes in patients with breast cancer. To determine whether STAT3 pathways were changed in the treatment groups, enrichment of JAKSTAT3 or IL-6 pathway-related gene signatures in the post-window phase samples compared to pre-window phase samples was analyzed. Enrichment analysis for JAK-STAT and IL-6 hallmark signatures were calculated using gene set variation analysis (GSVA) package. Each hospital followed their institutional guidelines for CRP and IL-6 measurements.
Time Frame: 28 weeks
Population: Subset (n=4, patients allocated to paclitaxel alone as neoadjuvant therapy; n=13, patients allocated to ruxolitinib plus paclitaxel given as neoadjuvant therapy) of the overall population allocated to neoadjuvant therapy (n=6; n=17, respectively) who had blood samples successfully assayed at both baseline and 28 wk timepoints.
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter
Arm/Group | Paclitaxel Alone Given As Neoadjuvant Therapy, After Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy
Number analyzed (Participants) | 4 | 13
picograms per milliliter | 0.3 [-0.1 to 4.0] | 1.6 [0.5 to 3.3]

9. Secondary Outcome: Changes in C-reactive Protein (CRP) Plasma Levels During Treatment
Description: Systemic biologic responses to ruxolitinib were assessed using serum IL-6 and c-reactive protein (CRP) levels. CRP levels are associated with poor prognosis and increased inflammatory response. Therefore, CRP levels in combination with pSTAT3 staining, could potentially be used as a more reliable method to select patients who would benefit from ruxolitinib treatment. To further analyze the effect of ruxolitinib throughout treatment, serum for CRP assessment was collected from patients at pre-window phase, post-window-phase, following 12-week neoadjuvant paclitaxel with or without ruxolitinib and immediately before surgery (pre-surgery). Each hospital followed their institutional guidelines for CRP measurements.
Time Frame: 28 weeks
Population: Subset (n=4, patients allocated to paclitaxel alone as neoadjuvant therapy; n=14, patients allocated to ruxolitinib plus paclitaxel given as neoadjuvant therapy) of the overall population allocated to neoadjuvant therapy (n=6; n=17, respectively) who had blood samples successfully assayed at both baseline and 28 wk timepoints.
Measure: Median (Inter-Quartile Range); unit: milligram per liter
Arm/Group | Paclitaxel Alone Given As Neoadjuvant Therapy, After Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy
Number analyzed (Participants) | 4 | 14
milligram per liter | -0.9 [-2.9 to 0.6] | 2.8 [-0.2 to 11.8]

ADVERSE EVENTS:
Time Frame: Deaths were assessed for 2 years and occurred during followup. Adverse Events were assessed for 28 weeks.
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 were utilized for adverse event reporting. A copy of the CTCAE version 4.0 can be downloaded from the CTEP website http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm.
Groups:
- Paclitaxel Alone Given As Neoadjuvant Therapy: Ruxolitinib alone (15 mg or 20 mg orally, depending on initial platelet count) is given in the run-in phase for 7 days. After the window phase, patients (n=6) who received ruxolitinib alone proceeded to neoadjuvant therapy with paclitaxel alone (80 mg/m2) for 12 weeks.
- Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy: After the run-in phase, patients (n=5) receiving single agent ruxolitinib (15 mg or 20 mg orally, depending on initial platelet count) twice daily for seven days, proceeded to neoadjuvant therapy with ruxolitinib plus paclitaxel for 12 weeks in addition to patients (n=12) who had received the combination of ruxolitinib plus paclitaxel (15 mg orally) twice daily for seven days in combination with one dose of paclitaxel (80 mg/m2; administered on day 1, denoted Cycle 0, Day 1) in the run-in phase, continued to receive the combination of ruxolitinib plus paclitaxel for a total of 12 weeks.
Arm/Group | Ruxolitinib Alone First | Ruxolitinib Plus Paclitaxel First | Paclitaxel Alone Given As Neoadjuvant Therapy | Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 3/6 | 5/17
Serious Adverse Events (participants affected / at risk) | 0/11 | 2/12 | 0/6 | 5/17
Other Adverse Events (participants affected / at risk) | 4/11 | 9/12 | 6/6 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib Alone First (N=11) | Ruxolitinib Plus Paclitaxel First (N=12) | Paclitaxel Alone Given As Neoadjuvant Therapy (N=6) | Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy (N=17)
Fatigue (General disorders) | 0 | 0 | 0 | 1 — General disorders and admin site conditions
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 2 | 0 | 0 — General disorders and administration site conditions
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib Alone First (N=11) | Ruxolitinib Plus Paclitaxel First (N=12) | Paclitaxel Alone Given As Neoadjuvant Therapy (N=6) | Ruxolitinib Plus Paclitaxel Given As Neoadjuvant Therapy (N=17)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 11
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 5 | 2 | 10
Chills (General disorders) | 0 | 0 | 0 | 2 — General disorders and admin site conditions
Edema face (General disorders) | 0 | 0 | 0 | 1 — General disorders and admin site conditions
Fatigue (General disorders) | 1 | 7 | 5 | 15 — General disorders and admin site conditions
Fever (General disorders) | 0 | 0 | 1 | 2 — General disorders and admin site conditions
Infusion related reaction (General disorders) | 0 | 0 | 1 | 0 — General disorders and admin site conditions
Pain (General disorders) | 0 | 0 | 0 | 3 — General disorders and admin site conditions
Skin infection (Infections and infestations) | 0 | 0 | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 3 | 6
White blood cell decreased (Investigations) | 0 | 0 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 5 | 8
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Skin/subcutaneous tissue disorders; Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 1 | 2
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT02876302/Prot_SAP_000.pdf